CLINICAL TRIAL: NCT00111800
Title: A 12-Week, Parallel-Group, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Dose Ranging Study to Evaluate the Efficacy, Safety and Tolerability of Denagliptin, Administered Orally, Once Daily, as Monotherapy in Subjects With Type 2 Diabetes Mellitus Followed by a 12-week Active Treatment Extension
Brief Title: A New Oral Treatment For Type II Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPB100925
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: NIDDM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Placebo (Placebo Comparator): Participants received oral dose of matching placebo capsule to denagliptin (DEN) once daily in the morning, 30 minutes (min) prior to breakfast during the main phase 12-weeks treatment period. Participants who were randomized to placebo in the main phase 12-weeks treatment period received oral dose of DEN 2.5 milligram (mg) once daily in the morning, 30 min prior to breakfast during the extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of placebo to the participants.
  Interventions: Drug: Placebo
- DEN 2.5 mg (Experimental): Participants received oral dose of DEN 2.5 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 2.5 mg to the participants.
  Interventions: Drug: DEN 2.5 mg
- DEN 7.5 mg (Experimental): Participants received oral dose of DEN 7.5 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 7.5 mg to the participants.
  Interventions: Drug: DEN 7.5 mg
- DEN 15 mg (Experimental): Participants received oral dose of DEN 15 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 15 mg to the participants.
  Interventions: Drug: DEN 15 mg
- DEN 30 mg (Experimental): Participants received oral dose of DEN 30 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 30 mg to the participants.
  Interventions: Drug: DEN 30 mg
- DEN 45 mg (Experimental): Participants received oral dose of DEN 45 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 45 mg to the participants.
  Interventions: Drug: DEN 45 mg

INTERVENTIONS:
Drug: Placebo — Placebo capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Arms: Placebo
Drug: DEN 2.5 mg — DEN 2.5 mg capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Other Names: GW823093 2.5 mg
  Arms: DEN 2.5 mg
Drug: DEN 7.5 mg — DEN 7.5 mg capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Other Names: GW823093 7.5 mg
  Arms: DEN 7.5 mg
Drug: DEN 15 mg — DEN 15 mg capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Other Names: GW823093 15 mg
  Arms: DEN 15 mg
Drug: DEN 30 mg — DEN 30 mg capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Other Names: GW823093 30 mg
  Arms: DEN 30 mg
Drug: DEN 45 mg — DEN 45 mg capsules which were white, opaque capsules with no identifying markings, containing white to off-white beads.
  Other Names: GW823093 45 mg
  Arms: DEN 45 mg

SUMMARY:
This is a 24-week study investigating the safety and efficacy of several dosages of a potential new oral medicine for Type II diabetes mellitus.

DETAILED DESCRIPTION:
A 12-Week, Parallel-Group, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Dose Ranging Study to Evaluate the Efficacy, Safety and Tolerability of GW823093, Administered Orally, Once Daily, as Monotherapy in Subjects With Type 2 Diabetes Mellitus followed by a 12-week Active Treatment Extension

ELIGIBILITY:
Inclusion criteria:

* Women must not be pregnant and must not be breastfeeding.
* Have Type II diabetes.
* Not taking any medicine for diabetes, or taking one oral medicine for their diabetes.

Exclusion criteria:

* Have any underlying or significant active disease that would prevent the subject from safely participating in the trial by the judgement of the study doctor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2005-04-28 (Actual); Primary Completion 2006-07-01 (Actual); Study Completion 2006-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (97):
- United States (35):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Pahrump, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Sewickley, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Vancouver, Washington
- Canada (11):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Cheb
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Třebíč
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Oulu
- Germany (26):
  - GSK Investigational Site, Bammental, Baden-Wurttemberg
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Königsfeld im Schwarzwald, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Stockach, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Bad Kreuznach, Hesse
  - GSK Investigational Site, Hirschhorn, Hesse
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Tostedt, Lower Saxony
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Lávrio
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- Latvia (5):
  - GSK Investigational Site, Jelgava
  - GSK Investigational Site, Ogre
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Talsi
  - GSK Investigational Site, Valmiera
- GSK Investigational Site, Ponce, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 28 April 2005 to 21 July 2006 across 94 centres from 9 countries.
Pre-assignment Details: A total of 375 participants received denagliptin ([DEN] 2.5, 7.5, 15, 30 or 45 milligram [mg]) or placebo which constituted the Safety Population. A total of 318 entered extension phase of study; 3 participants completed main phase but did not enter extension phase.
Groups:
- Placebo: Participants received oral dose of matching placebo capsule to DEN once daily in the morning, 30 minutes (min) prior to breakfast during the main phase 12-weeks treatment period. Participants who were randomized to placebo in the main phase 12-weeks treatment period received oral dose of DEN 2.5 mg once daily in the morning, 30 min prior to breakfast during the extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of placebo to the participants.
Period: Period 1: Main Phase (12 Weeks)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Started | 64 | 61 | 63 | 66 | 60 | 61
Completed | 49 | 47 | 54 | 60 | 55 | 56
Not Completed | 15 | 14 | 9 | 6 | 5 | 5
Not completed — Adverse Event | 5 | 4 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 2 | 4 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 0 | 0 | 1
Not completed — Lack of Efficacy | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Insufficient therapeutic effect | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Not meet treatment eligibility criteria | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Lack of glycaemic control | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Discontinued for not receiving incentive | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Would have been a drop out at Visit 4 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Fasting plasma glucose (FPG) below 140 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Elevated triglycerides | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Decrease in hemoglobin and hematocrit | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other-Protocol violator | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant went on extended holiday | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant's study medication stolen | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant moved out of area | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor requested withdrawal | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2: Extension Phase (12 Weeks)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Started | 48 | 47 | 54 | 59 | 55 | 55
Completed | 46 | 40 | 47 | 54 | 51 | 53
Not Completed | 2 | 7 | 7 | 5 | 4 | 2
Not completed — Adverse Event | 0 | 2 | 1 | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0 | 3 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1 | 0 | 1
Not completed — Insufficient therapeutic effect | 1 | 1 | 0 | 1 | 1 | 1
Not completed — Lack of Glycaemic Control | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Electrocardiogram (ECG) results | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant received metformin | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received oral dose of matching placebo capsule to DEN once daily in the morning, 30 min prior to breakfast during the main phase 12-weeks treatment period. Participants who were randomized to placebo in the main phase 12-weeks treatment period received oral dose of DEN 2.5 mg once daily in the morning, 30 min prior to breakfast during the extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of placebo to the participants.
- Total: Total of all reporting groups
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg | Total
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61 | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (10.89) | 58.6 (9.54) | 60.4 (12.41) | 59.9 (7.97) | 58.8 (9.95) | 59.2 (7.85) | 59.6 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 32 | 33 | 31 | 32 | 191
  Male | 32 | 30 | 31 | 33 | 29 | 29 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 1 | 6 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 5 | 2 | 5 | 3 | 1 | 4 | 20
  White | 57 | 58 | 57 | 60 | 53 | 55 | 340
  More than one race | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c is used to show in participants with diabetes, how well their diabetes is being controlled. The HbA1c test gives the average blood glucose levels over the pervious two to three months. The sample for HbA1c assessment was collected at Visit 5 (Week 0) and Visit 12 (Week 12). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 12) value. Analysis of covariance (ANCOVA) model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and Baseline measurement (continuous covariate). Last observation carried forward (LOCF) dataset defined as carrying forward of the last valid observation recorded on-treatment (scheduled or unscheduled) for participants who withdrew from the study to all remaining main phase visits was used. Adjusted mean is reported as least square (LS) mean.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent-to Treat (ITT) Population was defined as all randomized participants who received at least one dose of randomized study medication, had a Baseline assessment and had at least one corresponding on-therapy (scheduled or unscheduled) efficacy assessment. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
Percentage of HbA1c | 0.46 (0.105) | 0.18 (0.107) | -0.07 (0.104) | 0.01 (0.102) | -0.34 (0.107) | -0.38 (0.105)
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.061, ANCOVA; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.58 to 0.01] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.53, 95% CI 2-sided [-0.82 to -0.24] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.74 to -0.16] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.80, 95% CI 2-sided [-1.09 to -0.50] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.13 to -0.55] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg

2. Secondary Outcome: Change From Baseline in HbA1c at Week 4, 8, 16, 20 and 24
Description: HbA1c is use d to show in participants with diabetes, how well their diabetes is being controlled. The HbA1c test gives the average blood glucose levels over the pervious two to three months. The sample for HbA1c assessment was collected at Visit 5 (Week 0), Visit 9 (Week 4), Visit 11 (Week 8), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 4, Week 8, Week 16, Week 20 and Week 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
Percentage of HbA1c
  Week 4: number analyzed (Participants) | 58 | 56 | 59 | 61 | 56 | 57
  Week 4 | 0.22 (0.672) | -0.01 (0.505) | -0.11 (0.586) | -0.05 (0.474) | -0.25 (0.436) | -0.32 (0.445)
  Week 8: number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
  Week 8 | 0.21 (1.019) | 0.13 (0.753) | -0.04 (0.789) | -0.04 (0.645) | -0.36 (0.653) | -0.41 (0.579)
  Week 16: number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
  Week 16 | 0.40 (1.146) | 0.14 (0.934) | -0.04 (0.926) | 0.05 (0.790) | -0.30 (0.968) | -0.36 (0.821)
  Week 20: number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
  Week 20 | 0.31 (1.171) | 0.22 (1.143) | 0.02 (1.032) | 0.12 (0.853) | -0.25 (0.960) | -0.35 (0.823)
  Week 24: number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
  Week 24 | 0.35 (1.252) | 0.21 (1.184) | 0.06 (1.095) | 0.16 (0.942) | -0.28 (0.994) | -0.30 (0.900)

3. Secondary Outcome: Change From Baseline in FPG at Week 12
Description: The glycemic assessment of FPG measures a participant's blood sugar level after fasting or not eating anything for at least eight hours (h). The samples of FPG was collected was collected at Visit 5 (Week 0) and Visit 12 (Week 12). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 12) value. ANCOVA model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and Baseline measurement (continuous covariate). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimole per liter (mmol/L)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
Millimole per liter (mmol/L) | 0.52 (0.273) | 0.11 (0.282) | -0.28 (0.272) | -0.07 (0.270) | -0.95 (0.281) | -0.71 (0.276)
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.306, ANCOVA; Mean Difference (Net) = -0.40, 95% CI 2-sided [-1.18 to 0.37] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.039, ANCOVA; Mean Difference (Net) = -0.80, 95% CI 2-sided [-1.56 to -0.04] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.130, ANCOVA; Mean Difference (Net) = -0.58, 95% CI 2-sided [-1.34 to 0.17] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -1.46, 95% CI 2-sided [-2.23 to -0.69] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -1.22, 95% CI 2-sided [-1.99 to -0.46] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg

4. Secondary Outcome: Change From Baseline in FPG at Week 1, 2, 3, 4, 6, 8, 13, 14, 15, 16, 20 and 24
Description: The glycemic assessment of FPG measures a participant's blood sugar level after fasting or not eating anything for at least eight h. The sample for FPG assessment was collected at Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 1, 2, 3, 4, 6, 8, 13, 14, 15, 16, 20 and 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
mmol/L
  Week 1: number analyzed (Participants) | 61 | 58 | 62 | 63 | 57 | 60
  Week 1 | 0.33 (1.247) | 0.18 (2.178) | -0.45 (1.462) | -0.11 (1.782) | -0.73 (1.088) | -0.71 (1.605)
  Week 2: number analyzed (Participants) | 62 | 58 | 62 | 63 | 57 | 60
  Week 2 | 0.35 (1.385) | 0.23 (2.113) | -0.30 (1.575) | -0.25 (1.460) | -0.66 (1.514) | -0.69 (2.043)
  Week 3: number analyzed (Participants) | 62 | 58 | 62 | 63 | 57 | 60
  Week 3 | 0.37 (1.442) | 0.19 (1.975) | -0.65 (1.814) | -0.28 (1.603) | -0.81 (1.591) | -0.89 (1.844)
  Week 4: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 4 | 0.16 (1.595) | 0.22 (2.005) | -0.52 (2.235) | -0.43 (1.548) | -1.21 (1.514) | -1.31 (1.764)
  Week 6: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 6 | 0.17 (1.507) | 0.21 (2.149) | -0.61 (2.139) | -0.28 (1.420) | -1.02 (1.657) | -0.81 (1.882)
  Week 8: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 8 | 0.39 (1.745) | 0.18 (1.996) | -0.50 (2.235) | -0.33 (1.593) | -0.86 (1.869) | -1.10 (1.801)
  Week 13: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 13 | 0.25 (2.228) | 0.28 (2.305) | -0.19 (2.226) | -0.21 (2.016) | -0.84 (2.175) | -0.96 (2.058)
  Week 14: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 14 | 0.34 (2.348) | 0.31 (2.444) | -0.35 (2.492) | -0.11 (1.821) | -0.73 (2.279) | -0.86 (2.087)
  Week 15: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 15 | 0.16 (1.906) | 0.34 (2.206) | -0.40 (2.334) | -0.29 (1.828) | -0.88 (1.904) | -0.89 (1.952)
  Week 16: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 16 | 0.16 (1.950) | 0.07 (2.381) | -0.25 (2.514) | -0.41 (1.910) | -0.98 (2.213) | -0.89 (2.121)
  Week 20: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 20 | 0.16 (1.934) | 0.39 (2.898) | -0.04 (2.549) | 0.09 (1.913) | -1.04 (2.038) | -0.81 (2.344)
  Week 24: number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
  Week 24 | 0.67 (2.543) | 0.53 (2.807) | -0.07 (3.003) | 0.22 (2.186) | -1.01 (2.122) | -0.60 (2.364)

5. Secondary Outcome: Number of Participants Who Were HbA1c Responders at Week 12
Description: HbA1c is used to show in participants with diabetes, how well their diabetes is being controlled. The HbA1c test gives the average blood glucose levels over the pervious two to three months. The responders were defined as HbA1c values of <=6.5%, <7% and HbA1c reduction of >=0.7%. Analysis was done based on a logistic regression model with terms included for treatment, gender, prior therapy and Baseline measurement.
Time Frame: Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 59 | 56 | 59 | 62 | 56 | 58
Participants
  HbA1c <=6.5% | 6 | 4 | 4 | 5 | 9 | 8
  HbA1c <7% | 11 | 9 | 12 | 9 | 14 | 14
  HbA1c reduction >=0.7% | 10 | 6 | 14 | 10 | 21 | 17
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for HbA1c <=6.5%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.909, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.21 to 3.95]
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for HbA1c <=6.5%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.852, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.27 to 4.92]
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for HbA1c <=6.5%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.795, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.30 to 4.83]
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for HbA1c <=6.5%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.135, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.74 to 9.77]
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for HbA1c <=6.5%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.085, Regression, Logistic; Odds Ratio (OR) = 3.24, 95% CI 2-sided [0.85 to 12.37]
Statistical Analysis 6: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for HbA1c <7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.866, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.36 to 3.36]
Statistical Analysis 7: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for HbA1c <7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.202, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.69 to 5.76]
Statistical Analysis 8: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for HbA1c <7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.941, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.35 to 3.13]
Statistical Analysis 9: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for HbA1c <7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.152, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.76 to 6.13]
Statistical Analysis 10: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for HbA1c <7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.11 to 9.52]
Statistical Analysis 11: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for HbA1c reduction >=0.7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.198, Regression, Logistic; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.14 to 1.50]
Statistical Analysis 12: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for HbA1c reduction >=0.7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.481, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.53 to 3.85]
Statistical Analysis 13: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for HbA1c reduction >=0.7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.991, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.36 to 2.78]
Statistical Analysis 14: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for HbA1c reduction >=0.7%. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 3.65, 95% CI 2-sided [1.41 to 9.48]
Statistical Analysis 15: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for HbA1c reduction >=0.7%. A closed test procedure was used,P an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.161, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.76 to 5.24]

6. Secondary Outcome: Number of Participants of FPG Responders at Week 12
Description: The glycemic assessment of FPG measures a participant's blood sugar level after fasting or not eating anything for at least eight h. The responders were defined as FPG value of <7 mmol/L and FPG reduction value of >=1.7 mmol/L. Analysis was done based on a logistic regression model with terms included for treatment, gender, prior therapy and Baseline measurement.
Time Frame: Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 58 | 62 | 63 | 58 | 60
Participants
  FPG <7 mmol/L | 5 | 8 | 9 | 4 | 6 | 9
  FPG reduction >=1.7 mmol/L | 8 | 12 | 13 | 10 | 18 | 18
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for FPG <7mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.380, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.50 to 6.30]
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for FPG <7mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.145, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.72 to 9.11]
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for FPG <7mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.906, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.26 to 4.62]
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for FPG <7mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.509, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.41 to 5.91]
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for FPG <7mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.077, Regression, Logistic; Odds Ratio (OR) = 3.14, 95% CI 2-sided [0.89 to 11.14]
Statistical Analysis 6: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for FPG reduction >=1.7 mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.254, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.63 to 5.72]
Statistical Analysis 7: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for FPG reduction >=1.7 mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.396, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.55 to 4.62]
Statistical Analysis 8: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for FPG reduction >=1.7 mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.590, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.45 to 4.00]
Statistical Analysis 9: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for FPG reduction >=1.7 mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.15 to 9.13]
Statistical Analysis 10: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for FPG reduction >=1.7 mmol/L. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 3.00, 95% CI 2-sided [1.08 to 8.30]

7. Secondary Outcome: Change From Baseline in Fructosamine at Week 12
Description: The sample for fructosamine (total and corrected protein) assessment was collected at Visit 5 (Week 0) and Visit 12 (Week 12). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 12) value. ANCOVA model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and Baseline measurement (continuous covariate). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micromole (µmol/L)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 55 | 53 | 61 | 62 | 57 | 58
Micromole (µmol/L) | 19.9 (5.44) | 5.0 (5.55) | -2.5 (5.16) | -9.3 (5.12) | -19.7 (5.34) | -19.0 (5.29)
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.057, ANCOVA; Mean Difference (Net) = -14.9, 95% CI [-30.2 to 0.5] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Net) = -22.4, 95% CI [-37.1 to -7.6] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -29.2, 95% CI [-43.9 to -14.5] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -39.6, 95% CI 2-sided [-54.6 to -24.6] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -38.9, 95% CI 2-sided [-53.8 to -23.9] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg

8. Secondary Outcome: Change From Baseline in Fructosamine at Weeks 4, 8, 16, 20 and 24
Description: The sample for fructosamine (total and corrected protein) assessment was collected at Visit 5 (Week 0), Visit 9 (Week 4), Visit 11 (Week 8), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 4, 8, 16, 20 and 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
µmol/L
  Week 4: number analyzed (Participants) | 53 | 53 | 58 | 61 | 54 | 56
  Week 4 | 10.3 (38.09) | -4.3 (37.01) | -2.9 (34.08) | -10.1 (33.64) | -14.8 (29.36) | -22.0 (36.58)
  Week 8: number analyzed (Participants) | 55 | 53 | 61 | 61 | 57 | 58
  Week 8 | 15.9 (49.33) | -2.1 (39.42) | -5.0 (31.93) | -7.7 (32.84) | -20.2 (34.06) | -23.6 (33.32)
  Week 16: number analyzed (Participants) | 55 | 53 | 61 | 62 | 57 | 58
  Week 16 | 8.2 (48.67) | -0.5 (48.06) | -3.0 (39.37) | -3.5 (45.02) | -12.8 (43.62) | -18.6 (39.53)
  Week 20: number analyzed (Participants) | 55 | 53 | 61 | 62 | 57 | 58
  Week 20 | 14.7 (54.10) | 3.3 (51.12) | 0.3 (39.36) | -2.0 (46.96) | -9.6 (47.49) | -17.3 (42.07)
  Week 24: number analyzed (Participants) | 55 | 53 | 61 | 62 | 57 | 58
  Week 24 | 11.6 (56.07) | 6.7 (53.75) | 7.1 (49.03) | 7.0 (47.77) | -11.0 (48.02) | -10.9 (41.81)

9. Secondary Outcome: Change From Baseline in Fasting Serum Insulin and Pro-insulin at Week 12
Description: The assessment of fasting serum insulin measures a participant's serum insulin level after fasting or not eating anything for at least eight h. The sample for fasting serum insulin and pro-insulin was collected at Visit 5 (Week 0) and Visit 12 (Week 12). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 12) value. ANCOVA model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and baseline measurement (continuous covariate). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Picomole (pmol)/L
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
Picomole (pmol)/L
  Fasting serum insulin: number analyzed (Participants) | 56 | 52 | 58 | 62 | 53 | 54
  Fasting serum insulin | -2.04 (8.514) | -10.55 (8.804) | 12.14 (8.355) | 5.27 (8.057) | 3.23 (8.732) | 10.70 (8.641)
  Pro-insulin: number analyzed (Participants) | 57 | 53 | 61 | 62 | 56 | 58
  Pro-insulin | -4.28 (2.332) | -0.97 (2.418) | -1.21 (2.248) | -4.63 (2.228) | -6.49 (2.348) | -1.53 (2.307)
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for fasting serum insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.489, ANCOVA; Mean Difference (Net) = -8.51, 95% CI 2-sided [-32.66 to 15.65] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg for fasting serum insulin
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for fasting serum insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.237, ANCOVA; Mean Difference (Net) = 14.18, 95% CI 2-sided [-9.37 to 37.72] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg for fasting serum insulin
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for fasting serum insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.534, ANCOVA; Mean Difference (Net) = 7.31, 95% CI [-15.79 to 30.42] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg for fasting serum insulin
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for fasting serum insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.665, ANCOVA; Mean Difference (Net) = 5.27, 95% CI 2-sided [-18.64 to 29.17] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg for fasting serum insulin
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for fasting serum insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.295, ANCOVA; Mean Difference (Net) = 12.74, 95% CI 2-sided [-11.18 to 36.65] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg for fasting serum insulin
Statistical Analysis 6: Comparison: Placebo vs DEN 2.5 mg; Placebo versus DEN 2.5 mg for pro-insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.327, ANCOVA; Mean Difference (Net) = 3.31, 95% CI 2-sided [-3.32 to 9.94] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg for pro-insulin
Statistical Analysis 7: Comparison: Placebo vs DEN 7.5 mg; Placebo versus DEN 7.5 mg for pro-insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.345, ANCOVA; Mean Difference (Net) = 3.06, 95% CI 2-sided [-3.31 to 9.44] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg for pro-insulin
Statistical Analysis 8: Comparison: Placebo vs DEN 15 mg; Placebo versus DEN 15 mg for pro-insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.914, ANCOVA; Mean Difference (Net) = -0.35, 95% CI 2-sided [-6.70 to 6.00] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg for pro-insulin
Statistical Analysis 9: Comparison: Placebo vs DEN 30 mg; Placebo versus DEN 30 mg for pro-insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.504, ANCOVA; Mean Difference (Net) = -2.21, 95% CI 2-sided [-8.71 to 4.29] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg for pro-insulin
Statistical Analysis 10: Comparison: Placebo vs DEN 45 mg; Placebo versus DEN 45 mg for pro-insulin. A closed test procedure was used, in an hierarchical manner, that is, test was applied sequentially where testing does not proceed to the next step unless the previous test was found to be significant; Test type: Superiority; p = 0.403, ANCOVA; Mean Difference (Net) = 2.75, 95% CI 2-sided [-3.71 to 9.22] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg for pro-insulin

10. Secondary Outcome: Change From Baseline in Fasting Serum Insulin at Weeks 4, 8, 16, 20, 24 and Pro-insulin at Weeks 4 and 8
Description: The assessment of fasting serum insulin measures a participant's serum insulin level after fasting or not eating anything for at least eight h. The sample for fasting serum insulin was collected at Visit 5 (Week 0) Visit 9 (Week 4), Visit 11 (Week 8), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). The sample for pro-insulin was collected at Visit 5 (Week 0), Visit 9 (Week 4) and Visit 11 (Week 8). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 4, 8, 16, 20 and 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
pmol/L
  Week 4, Fasting serum insulin: number analyzed (Participants) | 53 | 51 | 55 | 61 | 49 | 52
  Week 4, Fasting serum insulin | 5.97 (50.769) | -3.83 (86.792) | 2.85 (75.790) | 1.67 (55.221) | 21.80 (78.596) | 7.23 (96.413)
  Week 8, Fasting serum insulin: number analyzed (Participants) | 56 | 52 | 58 | 61 | 53 | 55
  Week 8, Fasting serum insulin | 1.10 (42.239) | -11.90 (81.300) | 5.12 (81.860) | 2.29 (44.507) | 24.27 (72.846) | 25.21 (246.250)
  Week 16, Fasting serum insulin: number analyzed (Participants) | 56 | 52 | 58 | 62 | 53 | 55
  Week 16, Fasting serum insulin | 3.96 (55.879) | -9.02 (87.664) | 20.68 (148.343) | 1.05 (56.293) | 11.11 (33.429) | 9.83 (108.783)
  Week 20, Fasting serum insulin: number analyzed (Participants) | 56 | 52 | 58 | 62 | 53 | 55
  Week 20, Fasting serum insulin | 9.89 (73.956) | -0.65 (96.114) | 22.79 (148.597) | 4.76 (57.217) | 11.56 (41.611) | 0.68 (50.704)
  Week 24, Fasting serum insulin: number analyzed (Participants) | 56 | 52 | 58 | 62 | 53 | 55
  Week 24, Fasting serum insulin | 6.35 (55.319) | -6.66 (85.054) | 23.47 (157.791) | 11.62 (73.917) | 8.07 (36.118) | 0.69 (61.090)
  Week 4, Pro-insulin: number analyzed (Participants) | 55 | 53 | 58 | 61 | 52 | 56
  Week 4, Pro-insulin | -1.36 (21.662) | -2.42 (15.774) | -1.38 (24.872) | -4.48 (19.604) | -4.33 (18.011) | -5.55 (20.885)
  Week 8, Pro-insulin: number analyzed (Participants) | 57 | 53 | 61 | 61 | 56 | 58
  Week 8, Pro-insulin | 0.00 (18.948) | -4.23 (16.204) | -3.48 (16.865) | -4.59 (18.539) | -3.88 (18.139) | -4.45 (26.313)

11. Secondary Outcome: Change From Baseline in Pro-insulin at Week 16, 20 and 24.
Description: The sample for pro-insulin was collected at Visit 5 (Week 0), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 16, 20 and 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: ITT Population without LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
pmol/L
  Week 16: number analyzed (Participants) | 44 | 40 | 51 | 55 | 51 | 52
  Week 16 | -2.32 (19.820) | -4.45 (20.161) | -3.27 (16.672) | -4.24 (25.786) | -4.67 (13.882) | -1.35 (33.282)
  Week 20: number analyzed (Participants) | 44 | 37 | 49 | 55 | 49 | 53
  Week 20 | -2.52 (11.898) | 1.11 (26.455) | -2.24 (17.156) | -4.95 (17.947) | -4.84 (20.063) | -2.23 (22.270)
  Week 24: number analyzed (Participants) | 44 | 36 | 48 | 54 | 49 | 47
  Week 24 | -3.61 (15.914) | -0.64 (21.485) | -0.65 (31.694) | -3.07 (23.950) | -4.47 (20.598) | -2.34 (22.484)

12. Secondary Outcome: Change From Baseline in Pro-insulin to Insulin Ratio at Week 12
Description: The samples for pro-insulin and insulin was collected at Visit 5 (Week 0) and Visit 12 (Week 12). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 12) value. ANCOVA model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and baseline measurement (continuous covariate). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 56 | 52 | 58 | 62 | 52 | 54
Ratio | -0.02 (0.018) | 0.01 (0.019) | -0.04 (0.018) | -0.06 (0.017) | -0.08 (0.018) | -0.06 (0.018)
Statistical Analysis 1: Comparison: Placebo vs DEN 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.286, ANCOVA; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.02 to 0.08] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 2.5 mg
Statistical Analysis 2: Comparison: Placebo vs DEN 7.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.457, ANCOVA; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.07 to 0.03] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 7.5 mg
Statistical Analysis 3: Comparison: Placebo vs DEN 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.136, ANCOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.09 to 0.01] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 15 mg
Statistical Analysis 4: Comparison: Placebo vs DEN 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.11 to -0.01] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 30 mg
Statistical Analysis 5: Comparison: Placebo vs DEN 45 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.094, ANCOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.09 to 0.01] — The point estimate was calculated as least square mean difference (net values) of placebo and DEN 45 mg

13. Secondary Outcome: Change From Baseline in Pro-insulin to Insulin Ratio at Week 4 and 8
Description: The samples for pro-insulin and insulin was collected at Visit 5 (Week 0), Visit 9 (Week 4) and Visit 11 (Week 8). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 4 and 8) values. ANCOVA model for analysis was used with the terms for gender, prior therapy (diet & exercise/monotherapy), treatment, region and baseline measurement (continuous covariate). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Week 0) and Week 4 and 8
Population: ITT Population with LOCF dataset was used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 59 | 62 | 63 | 58 | 60
Ratio
  Week 4: number analyzed (Participants) | 53 | 51 | 55 | 61 | 48 | 52
  Week 4 | -0.02 (0.197) | -0.03 (0.176) | -0.03 (0.137) | -0.07 (0.169) | -0.13 (0.146) | -0.05 (0.137)
  Week 8: number analyzed (Participants) | 56 | 52 | 58 | 61 | 52 | 54
  Week 8 | 0.02 (0.133) | -0.01 (0.229) | -0.05 (0.120) | -0.07 (0.177) | -0.11 (0.174) | -0.07 (0.150)

14. Secondary Outcome: Number of Participants With Any Adverse Events (AE) or Serious Adverse Events (SAE) and Events of Hypoglycaemia
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. Medications that lowered blood glucose were capable of producing hypoglycemia or symptoms of hypoglycemia. Participants were provided with a hypoglycemic symptoms log at each visit and were asked to record symptoms of hypoglycemia.
Time Frame: Up to Week 25
Population: Safety population was defined as all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Participants
  Any AE | 28 | 26 | 31 | 36 | 29 | 30
  Any SAE | 1 | 1 | 2 | 0 | 4 | 3
  Any event of hypoglycaemia | 2 | 0 | 0 | 2 | 0 | 0

15. Secondary Outcome: Number of Participants With AE and Event of Hypoglycaemia of Mild, Moderate and Severe
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Medications that lowered blood glucose were capable of producing hypoglycemia or symptoms of hypoglycemia. Participants were provided with a hypoglycemic symptoms log at each visit and were asked to record symptoms of hypoglycemia. The assessment of severity was done by the investigator. A mild AE was defined as an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities. A moderate AE was defined as an event that was sufficiently discomforting to interfere with normal everyday activities. A severe AE was defined as an event that prevents normal everyday activities.
Time Frame: Up to Week 25
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Participants
  AE-Mild | 16 | 7 | 21 | 14 | 9 | 14
  AE-Moderate | 12 | 14 | 9 | 21 | 17 | 11
  AE-Severe | 0 | 5 | 1 | 1 | 3 | 5
  Hypoglycaemia-Mild | 2 | 0 | 0 | 2 | 0 | 0
  Hypoglycaemia-Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycaemia-Severe | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Change From Baseline Value of Potential Clinical Concern (PCC) in Vital Signs at Any Time During Therapy
Description: The vital sign assessments include systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR). The assessments were done pre-dose at Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week 1 to 24) values. The criteria for PCC included: HR increase or decrease from Baseline >30 beats per minute (bpm) and <50 or >120 bpm; SBP increase or decrease from Baseline >30 millimeter of mercury (mmHg) in the same posture and >170 or <100 mmHg; increase or decrease from Baseline >20 mmHg in same posture and >110 or <50 mmHg.
Time Frame: Baseline (Week 0) up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- DEN 30 mg: Participants received oral dose of DEN 15 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 15 mg to the participants.
- DEN 15 mg: Participants received oral dose of DEN 30 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 30 mg to the participants.
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 30 mg | DEN 15 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 60 | 62 | 63 | 59 | 60
Participants
  SBP, High | 4 | 4 | 1 | 5 | 4 | 6
  SBP, Low | 4 | 3 | 2 | 4 | 4 | 1
  DBP, High | 3 | 2 | 3 | 2 | 3 | 2
  DBP, Low | 3 | 3 | 2 | 4 | 1 | 3
  HR, High | 1 | 0 | 1 | 0 | 3 | 0
  HR, Low | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Body Weight Over Time
Description: The assessment of body weight was done during the run-in phase, randomized treatment phase and Follow-up at Visit 2 (Week -5), Visit 3 (Week -4), Visit 4 (Week -2), Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20), Visit 12 (Week 12), Visit 18 (Week 24) and Visit 19 (Week 25). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week -5 to 24) values.
Time Frame: Baseline (Week 0) and Week -5 to 25 (Follow-up)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Groups:
- DEN 2.5 mg: Participants received oral dose of matching placebo capsule to DEN once daily in the morning, 30 min prior to breakfast during the main phase 12-weeks treatment period. Participants who were randomized to placebo in the main phase 12-weeks treatment period received oral dose of DEN 2.5 mg once daily in the morning, 30 min prior to breakfast during the extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of placebo to the participants.
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Kilogram (kg)
  Week -5: number analyzed (Participants) | 64 | 61 | 62 | 63 | 60 | 61
  Week -5 | 1.09 (2.138) | 0.94 (1.923) | 0.52 (1.321) | 0.53 (1.740) | 1.24 (1.922) | 0.63 (1.808)
  Week -4: number analyzed (Participants) | 64 | 61 | 62 | 63 | 60 | 61
  Week -4 | 0.64 (1.624) | 0.83 (1.625) | 0.25 (1.178) | 0.23 (1.396) | 0.79 (1.676) | 0.58 (1.329)
  Week -2: number analyzed (Participants) | 63 | 61 | 59 | 63 | 59 | 61
  Week -2 | 0.31 (1.680) | 0.64 (1.175) | 0.12 (0.895) | 0.01 (1.167) | 0.35 (1.529) | 0.20 (0.894)
  Week 1: number analyzed (Participants) | 61 | 60 | 62 | 63 | 58 | 60
  Week 1 | -0.06 (1.547) | -0.10 (0.927) | -0.06 (0.928) | 0.10 (0.818) | 0.22 (1.396) | 0.09 (1.023)
  Week 2: number analyzed (Participants) | 60 | 58 | 60 | 63 | 57 | 60
  Week 2 | -0.25 (1.687) | 0.05 (1.935) | -0.26 (1.085) | -0.24 (1.060) | -0.34 (2.253) | -0.21 (1.264)
  Week 3: number analyzed (Participants) | 55 | 58 | 59 | 61 | 57 | 57
  Week 3 | -0.25 (1.724) | -0.38 (1.458) | -0.32 (1.135) | -0.25 (1.266) | -0.31 (1.364) | -0.21 (1.625)
  Week 4: number analyzed (Participants) | 57 | 56 | 58 | 60 | 58 | 58
  Week 4 | -0.22 (1.761) | -0.47 (1.730) | -0.42 (1.210) | -0.28 (1.386) | -0.60 (1.448) | 0.10 (1.722)
  Week 6: number analyzed (Participants) | 54 | 51 | 57 | 60 | 57 | 55
  Week 6 | -0.47 (1.394) | -0.65 (2.413) | -0.34 (1.413) | -0.30 (1.601) | -0.68 (2.070) | -0.29 (2.285)
  Week 8: number analyzed (Participants) | 52 | 49 | 56 | 60 | 57 | 56
  Week 8 | -0.42 (2.023) | -0.82 (2.743) | -0.38 (1.817) | -0.25 (1.450) | -0.56 (2.213) | -0.48 (2.435)
  Week 12: number analyzed (Participants) | 49 | 48 | 55 | 60 | 56 | 56
  Week 12 | -0.78 (2.332) | -0.96 (2.869) | -0.71 (1.885) | -0.36 (2.009) | -0.51 (2.745) | -0.50 (2.422)
  Week 13: number analyzed (Participants) | 47 | 47 | 54 | 57 | 52 | 53
  Week 13 | -0.93 (2.435) | -1.01 (3.105) | -0.68 (1.988) | -0.20 (1.971) | -0.35 (2.761) | -0.26 (2.617)
  Week 14: number analyzed (Participants) | 44 | 46 | 52 | 55 | 53 | 53
  Week 14 | -0.87 (2.279) | -1.13 (3.304) | -0.52 (2.012) | -0.06 (2.060) | -0.11 (2.781) | -0.46 (2.513)
  Week 15: number analyzed (Participants) | 45 | 44 | 53 | 56 | 53 | 55
  Week 15 | -1.06 (2.540) | -1.34 (3.019) | -0.72 (2.072) | -0.05 (2.186) | -0.24 (2.991) | -0.31 (2.587)
  Week 16: number analyzed (Participants) | 46 | 43 | 52 | 56 | 53 | 55
  Week 16 | -0.86 (2.836) | -1.36 (3.222) | -0.56 (1.920) | -0.31 (2.428) | -0.56 (3.144) | -0.45 (2.471)
  Week 20: number analyzed (Participants) | 46 | 41 | 50 | 55 | 51 | 55
  Week 20 | -0.89 (3.002) | -1.42 (3.604) | -0.59 (2.225) | -0.07 (2.666) | -0.30 (3.275) | -0.49 (2.628)
  Week 24: number analyzed (Participants) | 46 | 40 | 48 | 54 | 51 | 53
  Week 24 | -1.35 (3.343) | -1.86 (3.996) | -0.24 (2.185) | -0.31 (3.195) | -0.82 (3.517) | -0.43 (2.879)
  Week 25: number analyzed (Participants) | 46 | 40 | 46 | 54 | 51 | 52
  Week 25 | -0.97 (3.207) | -1.56 (3.558) | -0.45 (2.264) | -0.13 (3.048) | -0.65 (3.492) | -0.33 (2.892)

18. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Over Time
Description: BMI is an estimated the body fat of the participants, based on body weight divided by height squared. Height was assessed at Screening (Visit 2, Week -5) and confirmed at Baseline (Visit 5, Week 0). Weight was assessed at all Visits (Visit -5 to Visit 19). BMI was calculated during the run-in phase, randomized treatment phase and Follow-up at Visit 2 (Week -5), Visit 3 (Week -4), Visit 4 (Week -2), Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20), Visit 12 (Week 12), Visit 18 (Week 24) and Visit 19 (Week 25). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week -5 to 24) values.
Time Frame: Baseline (Week 0) and Week -5 to 25 (Follow-up)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: kg/meter square (m^2)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
kg/meter square (m^2)
  Week -5: number analyzed (Participants) | 64 | 61 | 62 | 63 | 60 | 61
  Week -5 | 0.374 (0.7989) | 0.392 (0.7566) | 0.183 (0.6269) | 0.207 (0.6319) | 0.538 (0.8620) | 0.239 (0.7085)
  Week -4: number analyzed (Participants) | 64 | 61 | 62 | 63 | 60 | 61
  Week -4 | 0.233 (0.6648) | 0.353 (0.7561) | 0.098 (0.5932) | 0.102 (0.5311) | 0.393 (0.8380) | 0.228 (0.5114)
  Week -2: number analyzed (Participants) | 63 | 61 | 59 | 63 | 59 | 61
  Week -2 | 0.108 (0.6859) | 0.292 (0.6340) | 0.029 (0.4579) | 0.015 (0.4473) | 0.231 (0.8162) | 0.090 (0.3338)
  Week 1: number analyzed (Participants) | 61 | 60 | 62 | 63 | 58 | 60
  Week 1 | -0.025 (0.5418) | -0.037 (0.3218) | -0.025 (0.3264) | 0.032 (0.2852) | 0.057 (0.4327) | 0.030 (0.3405)
  Week 2: number analyzed (Participants) | 60 | 58 | 60 | 63 | 57 | 60
  Week 2 | -0.091 (0.5994) | 0.015 (0.6716) | -0.089 (0.3943) | -0.091 (0.3694) | -0.130 (0.7748) | -0.077 (0.4441)
  Week 3: number analyzed (Participants) | 55 | 58 | 59 | 61 | 57 | 57
  Week 3 | -0.090 (0.6028) | -0.131 (0.4948) | -0.111 (0.3975) | -0.095 (0.4416) | -0.112 (0.4597) | -0.069 (0.5451)
  Week 4: number analyzed (Participants) | 57 | 56 | 58 | 60 | 58 | 58
  Week 4 | -0.076 (0.6281) | -0.169 (0.5870) | -0.140 (0.4301) | -0.094 (0.4858) | -0.218 (0.5059) | 0.035 (0.6149)
  Week 6: number analyzed (Participants) | 54 | 51 | 57 | 60 | 57 | 55
  Week 6 | -0.165 (0.4784) | -0.237 (0.8112) | -0.118 (0.5153) | -0.107 (0.5504) | -0.243 (0.7277) | -0.103 (0.8156)
  Week 8: number analyzed (Participants) | 52 | 49 | 56 | 60 | 57 | 56
  Week 8 | -0.158 (0.7015) | -0.303 (0.9424) | -0.128 (0.6772) | -0.080 (0.4984) | -0.211 (0.7819) | -0.173 (0.8603)
  Week 12: number analyzed (Participants) | 49 | 48 | 55 | 60 | 56 | 56
  Week 12 | -0.282 (0.8331) | -0.356 (0.9912) | -0.247 (0.6796) | -0.127 (0.7081) | -0.195 (0.9608) | -0.179 (0.8777)
  Week 13: number analyzed (Participants) | 47 | 47 | 54 | 57 | 52 | 53
  Week 13 | -0.324 (0.8814) | -0.377 (1.0859) | -0.238 (0.7310) | -0.064 (0.6939) | -0.157 (1.0077) | -0.083 (0.9680)
  Week 14: number analyzed (Participants) | 44 | 46 | 52 | 55 | 53 | 53
  Week 14 | -0.311 (0.7919) | -0.421 (1.1495) | -0.189 (0.7403) | -0.014 (0.7241) | -0.074 (1.0056) | -0.150 (0.9222)
  Week 15: number analyzed (Participants) | 45 | 44 | 53 | 56 | 53 | 55
  Week 15 | -0.375 (0.8965) | -0.485 (1.0575) | -0.255 (0.7621) | -0.006 (0.7797) | -0.111 (1.0993) | -0.103 (0.9438)
  Week 16: number analyzed (Participants) | 46 | 43 | 52 | 56 | 53 | 55
  Week 16 | -0.306 (1.0187) | -0.494 (1.1385) | -0.200 (0.7002) | -0.106 (0.8592) | -0.215 (1.1414) | -0.147 (0.8926)
  Week 20: number analyzed (Participants) | 46 | 41 | 50 | 55 | 51 | 55
  Week 20 | -0.312 (1.0837) | -0.524 (1.2742) | -0.211 (0.8145) | -0.015 (0.9340) | -0.138 (1.1961) | -0.171 (0.9598)
  Week 24: number analyzed (Participants) | 46 | 40 | 48 | 54 | 51 | 53
  Week 24 | -0.494 (1.1899) | -0.672 (1.4019) | -0.080 (0.7930) | -0.105 (1.1095) | -0.341 (1.2751) | -0.146 (1.0313)
  Week 25: number analyzed (Participants) | 46 | 40 | 46 | 54 | 51 | 52
  Week 25 | -0.350 (1.1468) | -0.571 (1.2553) | -0.152 (0.8295) | -0.041 (1.0595) | -0.268 (1.2877) | -0.107 (1.0426)

19. Secondary Outcome: Change From Baseline in Waist Circumference and Hip Circumference Over Time
Description: Waist and hip measurements were done at Screening (Visit 2, Week -5), Visit 5 (Week 0), Visit 12 (Week 12) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week -5 to 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Centimeter (cm)
  Hip circumference, Week -5: number analyzed (Participants) | 63 | 60 | 61 | 63 | 60 | 60
  Hip circumference, Week -5 | -0.1 (5.55) | 0.0 (4.49) | -0.5 (4.05) | -0.3 (3.92) | 0.6 (5.31) | -0.2 (4.61)
  Hip circumference, Week 12: number analyzed (Participants) | 48 | 48 | 53 | 58 | 53 | 56
  Hip circumference, Week 12 | -0.4 (4.73) | -0.5 (4.36) | -0.2 (3.25) | 0.6 (3.82) | -0.1 (4.77) | -2.6 (6.25)
  Hip circumference, Week 24: number analyzed (Participants) | 46 | 40 | 48 | 52 | 50 | 53
  Hip circumference, Week 24 | -1.6 (4.37) | -2.7 (5.37) | -0.3 (4.47) | 0.0 (5.11) | -0.9 (6.03) | -1.1 (3.67)
  Waist circumference, Week -5: number analyzed (Participants) | 63 | 60 | 62 | 63 | 60 | 60
  Waist circumference, Week -5 | 1.0 (4.49) | 2.6 (4.19) | 0.9 (4.46) | 0.9 (5.16) | -1.4 (4.97) | 1.3 (6.08)
  Waist circumference, Week 12: number analyzed (Participants) | 48 | 48 | 53 | 58 | 53 | 56
  Waist circumference, Week 12 | -1.1 (4.90) | -0.5 (4.47) | -1.0 (3.26) | -0.4 (3.39) | -0.1 (4.78) | 1.2 (7.60)
  Waist circumference, Week 24: number analyzed (Participants) | 46 | 40 | 48 | 52 | 50 | 53
  Waist circumference, Week 24 | -1.9 (4.84) | -1.0 (5.38) | -0.9 (3.91) | 0.3 (4.80) | -1.1 (7.13) | -0.8 (5.70)

20. Secondary Outcome: Mean Change From Baseline in Waist to Hip Ratio Over Time
Description: Waist to hip ratio calculation from the waist and hip measurements were done at Screening (Visit 2, Week -5), Visit 5 (Week 0), Visit 12 (Week 12) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week -5 to 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Ratio
  Week -5: number analyzed (Participants) | 63 | 60 | 61 | 63 | 60 | 60
  Week -5 | 0.01 (0.086) | 0.02 (0.063) | 0.01 (0.063) | 0.01 (0.067) | -0.02 (0.060) | 0.01 (0.086)
  Week 12: number analyzed (Participants) | 48 | 48 | 53 | 58 | 53 | 56
  Week 12 | -0.01 (0.054) | -0.00 (0.070) | -0.01 (0.037) | -0.01 (0.047) | -0.00 (0.067) | 0.03 (0.109)
  Week 24: number analyzed (Participants) | 46 | 40 | 48 | 52 | 50 | 53
  Week 24 | -0.00 (0.054) | 0.01 (0.064) | -0.01 (0.039) | 0.00 (0.064) | -0.00 (0.083) | 0.00 (0.051)

21. Secondary Outcome: Change From Baseline in 12-lead ECG Over Time
Description: 12-lead ECGs were obtained during the study using an ECG machine that automatically calculated the HR and measured PR, QRS, RR, QT, and QTc intervals. The mean PR interval, RR interval, QRS duration, uncorrected QT interval (UncQT) and QTcB (QT corrected by Bazett's formula) and QTcF (corrected by Friedericia's formula) was calculated from automated ECG readings. ECG was read centrally and locally at Visit 2 (Week -5), Visit 5 (Week 0), Visit 9 (Week 4), Visit 12 (Week 12), Visit 16 (Week 16) and Visit 18 (Week 24). Baseline value was defined as the assessment done at Week 0. The change from Baseline was calculated by subtracting the Baseline value (Week 0) from the individual post-Baseline (Week -5 to 24) values.
Time Frame: Baseline (Week 0) up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Milliseconds (msec)
  PR interval, Week -5: number analyzed (Participants) | 56 | 56 | 57 | 57 | 58 | 58
  PR interval, Week -5 | -1.5 (13.52) | 1.0 (11.38) | 0.3 (13.59) | -0.1 (13.16) | -1.3 (13.42) | 0.4 (14.31)
  PR interval, Week 4: number analyzed (Participants) | 54 | 55 | 55 | 58 | 54 | 55
  PR interval, Week 4 | 1.4 (13.56) | 0.3 (13.03) | -1.1 (17.22) | -0.3 (14.05) | 0.5 (14.18) | -3.5 (22.94)
  PR interval, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  PR interval, Week 12 | -0.6 (14.18) | -0.4 (17.29) | -1.4 (14.67) | 1.7 (13.56) | 1.1 (14.19) | -4.1 (23.38)
  PR interval, Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  PR interval, Week 16 | 1.4 (14.80) | 0.4 (13.38) | 0.0 (14.24) | 1.0 (12.91) | 1.1 (13.07) | -2.4 (20.76)
  PR interval, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  PR interval, Week 24 | -0.2 (15.39) | -0.6 (11.79) | -1.5 (14.61) | 0.3 (12.11) | 1.4 (13.17) | -5.5 (21.87)
  QRS duration, Week -5: number analyzed (Participants) | 57 | 56 | 58 | 57 | 58 | 59
  QRS duration, Week -5 | -0.4 (8.22) | -1.4 (7.36) | 2.1 (8.21) | 1.0 (10.92) | -0.6 (7.80) | 1.4 (8.65)
  QRS duration, Week 4: number analyzed (Participants) | 55 | 55 | 55 | 58 | 54 | 55
  QRS duration, Week 4 | -2.0 (7.87) | -0.1 (7.84) | -0.5 (8.49) | 0.7 (10.35) | -0.6 (7.40) | 0.8 (8.36)
  QRS duration, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  QRS duration, Week 12 | -1.2 (7.26) | -0.2 (6.85) | 2.2 (8.65) | -0.1 (12.10) | 0.1 (7.29) | 0.9 (8.97)
  QRS duration, Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  QRS duration, Week 16 | -1.9 (8.28) | -1.4 (7.64) | 0.1 (8.68) | -1.1 (11.46) | -0.5 (7.56) | -0.8 (9.39)
  QRS duration, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  QRS duration, Week 24 | -2.4 (9.48) | -1.3 (8.29) | 1.5 (8.29) | 0.0 (12.13) | 0.8 (10.09) | -1.1 (8.33)
  UncQT, Week -5: number analyzed (Participants) | 57 | 56 | 58 | 57 | 58 | 59
  UncQT, Week -5 | -7.2 (20.58) | -6.6 (21.32) | -1.1 (21.36) | -5.7 (16.47) | -6.2 (20.34) | 1.6 (19.27)
  UncQT, Week 4: number analyzed (Participants) | 55 | 55 | 55 | 58 | 54 | 55
  UncQT, Week 4 | -4.7 (22.21) | -0.9 (18.52) | 0.4 (20.89) | 0.4 (18.28) | -0.6 (21.32) | 9.0 (18.34)
  UncQT, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  UncQT, Week 12 | -5.1 (20.62) | -6.7 (21.53) | -2.1 (19.20) | -3.5 (18.34) | -3.1 (17.18) | 0.2 (20.74)
  UncQT, Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  UncQT, Week 16 | -4.6 (23.44) | -1.7 (19.94) | 1.8 (20.28) | -0.3 (20.48) | -2.9 (20.11) | 1.5 (23.05)
  UncQT, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  UncQT, Week 24 | -4.0 (21.76) | -5.7 (22.50) | 1.2 (21.42) | -4.0 (19.52) | -1.3 (21.30) | 4.3 (19.99)
  QTcB interval, Week -5: number analyzed (Participants) | 57 | 56 | 58 | 57 | 58 | 59
  QTcB interval, Week -5 | -1.9 (20.79) | -0.8 (17.21) | -0.4 (19.51) | -3.6 (14.95) | -0.7 (18.37) | -0.7 (19.55)
  QTcB interval, Week 4: number analyzed (Participants) | 55 | 55 | 55 | 58 | 54 | 55
  QTcB interval, Week 4 | -6.8 (19.85) | -6.5 (15.93) | -1.1 (20.65) | -2.8 (15.10) | 3.4 (17.15) | 2.7 (17.44)
  QTcB interval, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  QTcB interval, Week 12 | -7.7 (22.46) | -4.2 (22.27) | -1.2 (18.28) | -2.8 (18.14) | 1.5 (17.86) | 0.0 (18.96)
  QTcB interval, Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  QTcB interval, Week 16 | -7.5 (21.52) | -2.1 (22.13) | -0.6 (23.84) | -2.5 (18.14) | 2.4 (20.20) | -0.3 (21.13)
  QTcB interval, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  QTcB interval, Week 24 | -5.4 (20.82) | -1.7 (17.94) | 1.3 (20.06) | -3.5 (21.66) | 1.9 (17.90) | -0.1 (17.55)
  QTcF interval, Week -5: number analyzed (Participants) | 57 | 56 | 58 | 57 | 58 | 59
  QTcF interval, Week -5 | -3.8 (18.10) | -3.0 (14.83) | -0.7 (17.28) | -4.4 (13.03) | -2.5 (15.28) | 0.2 (15.97)
  QTcF interval, Week 4: number analyzed (Participants) | 55 | 55 | 55 | 58 | 54 | 55
  QTcF interval, Week 4 | -6.1 (17.19) | -4.6 (13.17) | -0.5 (17.66) | -1.8 (13.06) | 2.1 (15.11) | 5.0 (13.05)
  QTcF interval, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  QTcF interval, Week 12 | -6.7 (18.74) | -5.1 (18.06) | -1.5 (15.42) | -3.2 (13.59) | -0.1 (13.35) | 0.1 (15.58)
  QTcF interval,Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  QTcF interval,Week 16 | -6.5 (17.67) | -2.2 (17.47) | 0.3 (19.10) | -1.9 (16.80) | 0.6 (16.97) | 0.4 (17.38)
  QTcF interval, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  QTcF interval, Week 24 | -5.0 (17.52) | -3.2 (15.93) | 1.3 (16.65) | -3.8 (18.73) | 0.8 (16.16) | 1.4 (13.67)
  RR interval, Week -5: number analyzed (Participants) | 57 | 56 | 58 | 57 | 58 | 59
  RR interval, Week -5 | -25.5 (91.91) | -22.7 (107.49) | -5.1 (100.41) | -9.7 (75.09) | -25.0 (101.94) | 9.3 (102.60)
  RR interval, Week 4: number analyzed (Participants) | 55 | 55 | 55 | 58 | 54 | 55
  RR interval, Week 4 | 10.8 (106.59) | 26.0 (99.73) | 4.7 (104.53) | 15.0 (88.09) | -17.5 (97.17) | 23.1 (105.94)
  RR interval, Week 12: number analyzed (Participants) | 46 | 45 | 51 | 59 | 53 | 52
  RR interval, Week 12 | 9.2 (103.33) | -5.6 (117.39) | -4.6 (102.36) | -3.1 (118.09) | -21.4 (103.46) | -2.2 (104.03)
  RR interval, Week 16: number analyzed (Participants) | 43 | 42 | 49 | 56 | 51 | 53
  RR interval, Week 16 | 13.3 (124.03) | 5.7 (115.66) | 10.9 (119.81) | 11.3 (82.95) | -24.4 (99.46) | 3.6 (121.42)
  RR interval, Week 24: number analyzed (Participants) | 43 | 39 | 46 | 51 | 50 | 50
  RR interval, Week 24 | 5.9 (109.76) | -13.4 (107.74) | -1.7 (119.94) | -2.7 (85.56) | -14.6 (97.99) | 17.2 (115.09)

22. Secondary Outcome: Number of Participants With Laboratory Clinical Chemistry Values of PCC at Any Time on Therapy
Description: The parameters of clinical chemistry included sodium, potassium, chloride, bicarbonate, lactate dehydrogenase ([LDH] if >2x upper limit of reference range, LDH isoenzymes were collected), total protein, albumin, blood urea nitrogen (BUN), creatinine, total bilirubin, direct bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), Calcium, phosphorus (inorganic) and uric acid. The assessments were done at Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Only those parameters for which at least one value of PCC was reported are summarized.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 60 | 62 | 63 | 59 | 60
Participants
  Albumin, High | 0 | 0 | 0 | 0 | 1 | 1
  AST, high | 0 | 0 | 0 | 0 | 1 | 0
  Calcium, Low | 3 | 5 | 5 | 3 | 3 | 10
  Carbon dioxide content/bicarbonate, low | 3 | 5 | 6 | 4 | 1 | 7
  Creatinine, high | 0 | 0 | 0 | 1 | 0 | 1
  Glucose, low | 0 | 0 | 1 | 1 | 0 | 1
  Phosphorus inorganic, high | 0 | 0 | 2 | 0 | 0 | 1
  Potassium,high | 11 | 4 | 8 | 7 | 7 | 10
  Sodium, high | 0 | 0 | 0 | 1 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0 | 2 | 2
  Total bilirubin, high | 2 | 2 | 1 | 1 | 2 | 1
  Uric scid, high | 0 | 0 | 1 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Laboratory Haematology Values of PCC at Any Time on Therapy
Description: The parameters of hematology included red blood cell (RBC) count, hemoglobin, hematocrit, platelet count and total white blood cell (WBC) count. The assessments were done at Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20) and Visit 18 (Week 24). Only those parameters for which at least one value of PCC was reported are summarized.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 62 | 60 | 62 | 63 | 59 | 60
Participants
  Hematocrit, high | 3 | 0 | 2 | 0 | 2 | 2
  Hematocrit, low | 1 | 4 | 0 | 1 | 0 | 1
  Hemoglobin, high | 3 | 1 | 3 | 0 | 1 | 2
  Hemoglobin, low | 1 | 3 | 1 | 0 | 1 | 0
  Platelet count, low | 0 | 0 | 0 | 0 | 1 | 0
  WBC count, high | 0 | 0 | 0 | 1 | 1 | 1

24. Secondary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Result
Description: The parameters of dipstick urinalysis included glucose, bilirubin, protein and ketones. The abnormal results of dispstick parameters were categorized for glucose as trace or 1/10 gram (g)/deciliter (dL %), 1+ or ¼ g/dL (%), 2+ or ½ g/dL (%), 3+ or 1 g/dL (%); for ketones as 1+ and trace; for proteins as 1+, 2+, 3+ and trace. The assessments were done at Visit 2 (Week -5), Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20), Visit 18 (Week 24) and Visit 19 (Week 25).
Time Frame: Up to Follow-up (Week 25)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Participants
  Week -5, Glucose, trace or 1/10 g/dL | 7 | 3 | 6 | 4 | 3 | 9
  Week -5, Glucose, 1+ or 1/4 g/dL | 3 | 6 | 4 | 3 | 5 | 2
  Week -5, Glucose, 2+ or 1/2 g/dL | 1 | 1 | 1 | 2 | 4 | 4
  Week -5, Glucose, 3+ or 1 g/dL | 5 | 3 | 3 | 1 | 4 | 3
  Week -5, Ketones, trace | 3 | 2 | 3 | 1 | 1 | 2
  Week -5, Ketones, 1+ | 1 | 1 | 1 | 0 | 0 | 0
  Week -5, Protein, trace | 8 | 4 | 9 | 5 | 5 | 3
  Week -5, Protein,1+ | 6 | 6 | 5 | 5 | 4 | 2
  Week -5, Protein, 2+ | 0 | 1 | 2 | 1 | 3 | 0
  Week -5, Protein, 3+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 0, Glucose, trace or 1/10 g/dL | 10 | 5 | 3 | 5 | 6 | 6
  Week 0, Glucose, 1+ or 1/4 g/dL | 3 | 5 | 7 | 7 | 2 | 5
  Week 0, Glucose, 2+ or 1/2 g/dL | 5 | 3 | 3 | 4 | 2 | 0
  Week 0, Glucose, 3+ or 1 g/dL | 3 | 6 | 5 | 4 | 2 | 8
  Week 0, Ketones, trace | 2 | 2 | 3 | 1 | 2 | 3
  Week 0, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 0, Protein, trace | 9 | 10 | 5 | 9 | 3 | 6
  Week 0, Protein,1+ | 8 | 2 | 4 | 4 | 5 | 2
  Week 0, Protein, 2+ | 1 | 1 | 2 | 3 | 2 | 0
  Week 0, Protein, 3+ | 0 | 1 | 0 | 0 | 0 | 0
  Week 1, Glucose, trace or 1/10 g/dL | 7 | 4 | 9 | 8 | 4 | 4
  Week 1, Glucose, 1+ or 1/4 g/dL | 5 | 7 | 3 | 3 | 2 | 4
  Week 1, Glucose, 2+ or 1/2 g/dL | 4 | 1 | 2 | 2 | 0 | 1
  Week 1, Glucose, 3+ or 1 g/dL | 6 | 7 | 5 | 1 | 1 | 5
  Week 1, Ketones, trace | 2 | 1 | 3 | 0 | 1 | 3
  Week 1, Ketones, 1+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 1, Protein, trace | 7 | 7 | 6 | 4 | 7 | 4
  Week 1, Protein,1+ | 7 | 6 | 2 | 3 | 2 | 0
  Week 1, Protein, 2+ | 0 | 0 | 1 | 1 | 1 | 0
  Week 1, Protein, 3+ | 0 | 0 | 1 | 0 | 0 | 0
  Week 2, Glucose, trace or 1/10 g/dL | 4 | 6 | 9 | 5 | 1 | 4
  Week 2, Glucose, 1+ or 1/4 g/dL | 1 | 3 | 2 | 1 | 7 | 5
  Week 2, Glucose, 2+ or 1/2 g/dL | 3 | 4 | 1 | 3 | 0 | 1
  Week 2, Glucose, 3+ or 1 g/dL | 7 | 8 | 6 | 3 | 0 | 3
  Week 2, Ketones, trace | 3 | 3 | 0 | 1 | 1 | 0
  Week 2, Ketones, 1+ | 1 | 0 | 1 | 0 | 0 | 0
  Week 2, Protein, trace | 4 | 5 | 6 | 6 | 5 | 4
  Week 2, Protein,1+ | 6 | 3 | 1 | 3 | 4 | 0
  Week 2, Protein, 2+ | 0 | 0 | 1 | 1 | 1 | 0
  Week 2, Protein, 3+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 3, Glucose, trace or 1/10 g/dL | 4 | 5 | 11 | 6 | 1 | 5
  Week 3, Glucose, 1+ or 1/4 g/dL | 3 | 7 | 2 | 2 | 2 | 2
  Week 3, Glucose, 2+ or 1/2 g/dL | 1 | 0 | 1 | 4 | 1 | 1
  Week 3, Glucose, 3+ or 1 g/dL | 8 | 7 | 2 | 3 | 2 | 4
  Week 3, Ketones, trace | 0 | 1 | 2 | 1 | 2 | 2
  Week 3, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 3, Protein, trace | 7 | 5 | 5 | 2 | 4 | 2
  Week 3, Protein, 1+ | 2 | 4 | 3 | 5 | 1 | 3
  Week 3, Protein, 2+ | 2 | 0 | 0 | 1 | 2 | 0
  Week 3, Protein, 3+ | 0 | 0 | 1 | 0 | 0 | 0
  Week 4, Glucose, trace or 1/10 g/dL | 3 | 8 | 5 | 7 | 3 | 4
  Week 4, Glucose, 1+ or 1/4 g/dL | 2 | 5 | 0 | 6 | 4 | 2
  Week 4, Glucose, 2+ or 1/2 g/dL | 1 | 5 | 3 | 1 | 2 | 4
  Week 4, Glucose, 3+ or 1 g/dL | 8 | 3 | 5 | 1 | 1 | 0
  Week 4, Ketones, trace | 1 | 1 | 1 | 1 | 0 | 0
  Week 4, Ketones, 1+ | 0 | 0 | 0 | 0 | 1 | 1
  Week 4, Protein, trace | 7 | 7 | 3 | 6 | 4 | 1
  Week 4, Protein, 1+ | 3 | 3 | 1 | 4 | 4 | 0
  Week 4, Protein, 2+ | 2 | 0 | 1 | 1 | 1 | 0
  Week 4, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 6, Glucose, trace or 1/10 g/dL | 6 | 7 | 5 | 9 | 6 | 3
  Week 6, Glucose, 1+ or 1/4 g/dL | 2 | 4 | 6 | 1 | 2 | 3
  Week 6, Glucose, 2+ or 1/2 g/dL | 4 | 5 | 2 | 1 | 1 | 1
  Week 6, Glucose, 3+ or 1 g/dL | 6 | 3 | 3 | 2 | 1 | 3
  Week 6, Ketones, trace | 2 | 1 | 2 | 1 | 0 | 2
  Week 6, Ketones, 1+ | 0 | 1 | 0 | 0 | 0 | 0
  Week 6, Protein, trace | 8 | 8 | 5 | 6 | 2 | 4
  Week 6, Protein, 1+ | 4 | 3 | 3 | 5 | 3 | 1
  Week 6, Protein, 2+ | 1 | 1 | 0 | 2 | 2 | 0
  Week 6, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 8, Glucose, trace or 1/10 g/dL | 6 | 5 | 5 | 7 | 3 | 5
  Week 8, Glucose, 1+ or 1/4 g/dL | 1 | 3 | 5 | 3 | 2 | 2
  Week 8, Glucose, 2+ or 1/2 g/dL | 2 | 2 | 2 | 5 | 2 | 3
  Week 8, Glucose, 3+ or 1 g/dL | 8 | 4 | 5 | 2 | 0 | 0
  Week 8, Ketones, trace | 1 | 1 | 0 | 0 | 3 | 1
  Week 8, Ketones, 1+ | 0 | 0 | 1 | 0 | 0 | 0
  Week 8, Protein, trace | 2 | 5 | 5 | 8 | 3 | 1
  Week 8, Protein, 1+ | 4 | 4 | 4 | 2 | 5 | 2
  Week 8, Protein, 2+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 8, Protein, 3+ | 0 | 0 | 0 | 1 | 0 | 0
  Week 12, Glucose, trace or 1/10 g/dL | 6 | 7 | 7 | 5 | 2 | 3
  Week 12, Glucose, 1+ or 1/4 g/dL | 1 | 6 | 2 | 2 | 1 | 6
  Week 12, Glucose, 2+ or 1/2 g/dL | 3 | 1 | 1 | 4 | 0 | 2
  Week 12, Glucose, 3+ or 1 g/dL | 6 | 6 | 7 | 2 | 1 | 0
  Week 12, Ketones, trace | 1 | 4 | 0 | 0 | 0 | 1
  Week 12, Ketones, 1+ | 0 | 1 | 0 | 0 | 0 | 0
  Week 12, Protein, trace | 7 | 6 | 5 | 6 | 4 | 4
  Week 12, Protein, 1+ | 1 | 5 | 3 | 4 | 4 | 0
  Week 12, Protein, 2+ | 1 | 0 | 0 | 0 | 1 | 0
  Week 12, Protein, 3+ | 0 | 0 | 0 | 1 | 0 | 0
  Week 13, Glucose, trace or 1/10 g/dL | 1 | 6 | 2 | 7 | 6 | 5
  Week 13, Glucose, 1+ or 1/4 g/dL | 2 | 1 | 1 | 7 | 1 | 4
  Week 13, Glucose, 2+ or 1/2 g/dL | 2 | 3 | 2 | 2 | 2 | 1
  Week 13, Glucose, 3+ or 1 g/dL | 7 | 6 | 6 | 1 | 1 | 2
  Week 13, Ketones, trace | 0 | 0 | 0 | 0 | 2 | 1
  Week 13, Ketones, 1+ | 0 | 0 | 1 | 0 | 0 | 0
  Week 13, Protein, trace | 3 | 6 | 0 | 4 | 8 | 3
  Week 13, Protein, 1+ | 2 | 2 | 4 | 3 | 1 | 1
  Week 13, Protein, 2+ | 1 | 0 | 0 | 1 | 2 | 0
  Week 13, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 14, Glucose, trace or 1/10 g/dL | 3 | 7 | 6 | 5 | 3 | 2
  Week 14, Glucose, 1+ or 1/4 g/dL | 0 | 5 | 3 | 3 | 0 | 2
  Week 14, Glucose, 2+ or 1/2 g/dL | 4 | 0 | 2 | 2 | 3 | 2
  Week 14, Glucose, 3+ or 1 g/dL | 7 | 3 | 3 | 1 | 1 | 3
  Week 14, Ketones, trace | 0 | 1 | 1 | 0 | 1 | 1
  Week 14, Ketones, 1+ | 0 | 0 | 0 | 0 | 1 | 0
  Week 14, Protein, trace | 2 | 3 | 3 | 3 | 3 | 4
  Week 14, Protein, 1+ | 3 | 3 | 4 | 3 | 4 | 1
  Week 14, Protein, 2+ | 0 | 0 | 1 | 1 | 1 | 0
  Week 14, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 15, Glucose, trace or 1/10 g/dL | 2 | 5 | 5 | 4 | 3 | 4
  Week 15, Glucose, 1+ or 1/4 g/dL | 5 | 4 | 3 | 5 | 2 | 1
  Week 15, Glucose, 2+ or 1/2 g/dL | 1 | 1 | 0 | 0 | 1 | 3
  Week 15, Glucose, 3+ or 1 g/dL | 6 | 4 | 5 | 2 | 1 | 2
  Week 15, Ketones, trace | 1 | 0 | 2 | 1 | 1 | 1
  Week 15, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 15, Protein, trace | 7 | 2 | 5 | 2 | 2 | 5
  Week 15, Protein, 1+ | 1 | 2 | 3 | 4 | 6 | 2
  Week 15, Protein, 2+ | 0 | 0 | 2 | 2 | 1 | 0
  Week 15, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 16, Glucose, trace or 1/10 g/dL | 7 | 4 | 4 | 5 | 0 | 6
  Week 16, Glucose, 1+ or 1/4 g/dL | 0 | 4 | 3 | 8 | 3 | 1
  Week 16, Glucose, 2+ or 1/2 g/dL | 2 | 0 | 3 | 0 | 1 | 3
  Week 16, Glucose, 3+ or 1 g/dL | 6 | 5 | 3 | 1 | 2 | 4
  Week 16, Ketones, trace | 2 | 1 | 0 | 1 | 0 | 1
  Week 16, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 16, Protein, trace | 2 | 1 | 4 | 1 | 5 | 3
  Week 16, Protein, 1+ | 2 | 3 | 4 | 4 | 1 | 3
  Week 16, Protein, 2+ | 0 | 0 | 1 | 1 | 0 | 0
  Week 16, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 20, Glucose, trace or 1/10 g/dL | 2 | 4 | 4 | 6 | 4 | 4
  Week 20, Glucose, 1+ or 1/4 g/dL | 2 | 1 | 3 | 3 | 5 | 4
  Week 20, Glucose, 2+ or 1/2 g/dL | 4 | 3 | 0 | 1 | 0 | 1
  Week 20, Glucose, 3+ or 1 g/dL | 3 | 4 | 4 | 3 | 2 | 4
  Week 20, Ketones, trace | 0 | 2 | 0 | 1 | 1 | 1
  Week 20, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 1
  Week 20, Protein, trace | 8 | 4 | 2 | 2 | 4 | 3
  Week 20, Protein, 1+ | 1 | 3 | 2 | 5 | 4 | 1
  Week 20, Protein, 2+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 20, Protein, 3+ | 0 | 0 | 0 | 1 | 0 | 0
  Week 24, Glucose, trace or 1/10 g/dL | 2 | 3 | 8 | 3 | 1 | 4
  Week 24, Glucose, 1+ or 1/4 g/dL | 1 | 5 | 2 | 7 | 1 | 1
  Week 24, Glucose, 2+ or 1/2 g/dL | 0 | 4 | 1 | 2 | 2 | 3
  Week 24, Glucose, 3+ or 1 g/dL | 7 | 1 | 3 | 5 | 2 | 1
  Week 24, Ketones, trace | 0 | 0 | 1 | 3 | 2 | 0
  Week 24, Ketones, 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 24, Protein, trace | 6 | 7 | 6 | 3 | 4 | 5
  Week 24, Protein, 1+ | 1 | 3 | 2 | 5 | 4 | 0
  Week 24, Protein, 2+ | 0 | 0 | 0 | 1 | 1 | 1
  Week 24, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Week 25, Glucose, trace or 1/10 g/dL | 7 | 3 | 9 | 4 | 0 | 6
  Week 25, Glucose, 1+ or 1/4 g/dL | 1 | 2 | 4 | 3 | 1 | 3
  Week 25, Glucose, 2+ or 1/2 g/dL | 3 | 0 | 2 | 4 | 1 | 0
  Week 25, Glucose, 3+ or 1 g/dL | 4 | 2 | 1 | 4 | 4 | 3
  Week 25, Ketones, trace | 2 | 0 | 1 | 0 | 0 | 0
  Week 25, Ketones, 1+ | 0 | 1 | 0 | 0 | 0 | 0
  Week 25, Protein, trace | 6 | 4 | 2 | 5 | 2 | 3
  Week 25, Protein, 1+ | 2 | 4 | 1 | 5 | 3 | 0
  Week 25, Protein, 2+ | 1 | 0 | 0 | 0 | 0 | 0
  Week 25, Protein, 3+ | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Urinalysis Microscopic Result
Description: The parameters of microscopic urinalysis included RBC and WBC. The microscopic urinalysis results for the parameters were categorized as cells of 0-1, 1-3, 3-5, 5-10, 10-15, 15-25, 25-50, 50-100 and innumerable. The assessments were done at Visit 2 (Week -5), Visit 5 (Week 0), Visit 6 (Week 1), Visit 7 (Week 2), Visit 8 (Week 3), Visit 9 (Week 4), Visit 10 (Week 6), Visit 11 (Week 8), Visit 12 (Week 12), Visit 13 (Week 13), Visit 14 (Week 14), Visit 15 (Week 15), Visit 16 (Week 16), Visit 17 (Week 20), Visit 18 (Week 24) and Visit 19 (Week 25).
Time Frame: Up to Follow-up (Week 25)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 64 | 61 | 63 | 66 | 60 | 61
Participants
  Week -5, RBC, 0-1 | 3 | 1 | 2 | 0 | 2 | 2
  Week -5, RBC, 1-3 | 3 | 4 | 1 | 2 | 2 | 1
  Week -5, RBC, 3-5 | 1 | 1 | 1 | 0 | 0 | 0
  Week -5, RBC, 5-10 | 2 | 3 | 0 | 0 | 2 | 1
  Week -5, RBC, 10-15 | 0 | 0 | 0 | 0 | 1 | 0
  Week -5, RBC, 15-25 | 0 | 0 | 0 | 0 | 0 | 1
  Week -5, RBC, ,25-50 | 1 | 0 | 0 | 0 | 0 | 0
  Week -5, RBC, 50-100 | 0 | 0 | 0 | 1 | 0 | 0
  Week -5, RBC, innumerable | 1 | 0 | 1 | 0 | 0 | 0
  Week -5, WBC, 0-1 | 7 | 4 | 3 | 1 | 3 | 1
  Week -5, WBC, 1-3 | 2 | 1 | 4 | 3 | 3 | 2
  Week -5, WBC, 3-5 | 2 | 2 | 1 | 0 | 3 | 2
  Week -5, WBC, 5-10 | 3 | 3 | 1 | 3 | 1 | 2
  Week -5, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week -5, WBC, 15-25 | 4 | 2 | 1 | 5 | 2 | 1
  Week -5, WBC, 25-50 | 2 | 1 | 1 | 2 | 4 | 1
  Week -5, WBC, 50-100 | 1 | 1 | 2 | 1 | 3 | 0
  Week -5, WBC, innumerable | 4 | 1 | 1 | 0 | 1 | 1
  Week 0, RBC, 0-1 | 3 | 0 | 3 | 1 | 0 | 0
  Week 0, RBC, 1-3 | 1 | 3 | 0 | 2 | 3 | 2
  Week 0, RBC, 3-5 | 3 | 4 | 0 | 0 | 1 | 1
  Week 0, RBC, 5-10 | 0 | 0 | 0 | 3 | 2 | 0
  Week 0, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0, RBC, 15-25 | 0 | 0 | 0 | 0 | 1 | 0
  Week 0, RBC, 25-50 | 1 | 0 | 2 | 0 | 1 | 0
  Week 0, RBC, 50-100 | 0 | 0 | 0 | 1 | 1 | 0
  Week 0, RBC, innumerable | 1 | 0 | 0 | 1 | 0 | 1
  Week 0, WBC, 0-1 | 6 | 2 | 4 | 3 | 2 | 2
  Week 0, WBC, 1-3 | 3 | 4 | 3 | 6 | 3 | 1
  Week 0, WBC, 3-5 | 4 | 4 | 0 | 1 | 2 | 0
  Week 0, WBC, 5-10 | 5 | 4 | 0 | 4 | 7 | 3
  Week 0, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0, WBC, 15-25 | 2 | 2 | 4 | 2 | 2 | 3
  Week 0, WBC, 25-50 | 0 | 4 | 5 | 2 | 4 | 1
  Week 0, WBC, 50-100 | 0 | 2 | 3 | 2 | 1 | 1
  Week 0, WBC, innumerable | 3 | 1 | 0 | 1 | 0 | 0
  Week 1, RBC, 0-1 | 2 | 1 | 2 | 2 | 0 | 1
  Week 1, RBC, 1-3 | 2 | 6 | 5 | 1 | 1 | 1
  Week 1, RBC, 3-5 | 2 | 1 | 0 | 2 | 0 | 1
  Week 1, RBC, 5-10 | 1 | 0 | 0 | 2 | 0 | 0
  Week 1, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1, RBC, 15-25 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1, RBC, 25-50 | 2 | 1 | 2 | 0 | 0 | 0
  Week 1, RBC, 50-100 | 1 | 0 | 1 | 0 | 1 | 1
  Week 1, RBC, innumerable | 0 | 0 | 0 | 1 | 0 | 0
  Week 1, WBC, 0-1 | 3 | 1 | 3 | 3 | 0 | 4
  Week 1, WBC, 1-3 | 6 | 6 | 6 | 5 | 2 | 0
  Week 1, WBC, 3-5 | 0 | 1 | 2 | 4 | 5 | 1
  Week 1, WBC, 5-10 | 4 | 2 | 3 | 2 | 1 | 1
  Week 1, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1, WBC, 15-25 | 3 | 0 | 3 | 1 | 1 | 2
  Week 1, WBC, 25-50 | 1 | 3 | 2 | 1 | 2 | 1
  Week 1, WBC, 50-100 | 3 | 1 | 4 | 1 | 4 | 2
  Week 1, WBC, innumerable | 1 | 1 | 0 | 0 | 2 | 0
  Week 2, RBC, 0-1 | 3 | 0 | 0 | 4 | 1 | 3
  Week 2, RBC, 1-3 | 3 | 3 | 0 | 1 | 4 | 2
  Week 2, RBC, 3-5 | 0 | 2 | 1 | 1 | 1 | 2
  Week 2, RBC, 5-10 | 1 | 0 | 0 | 0 | 0 | 3
  Week 2, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2, RBC, 15-25 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2, RBC, 25-50 | 3 | 1 | 1 | 3 | 0 | 0
  Week 2, RBC, 50-100 | 2 | 0 | 0 | 0 | 0 | 0
  Week 2, RBC, innumerable | 0 | 0 | 0 | 0 | 0 | 0
  Week 2, WBC, 0-1 | 3 | 1 | 2 | 0 | 3 | 6
  Week 2, WBC, 1-3 | 6 | 3 | 2 | 2 | 3 | 0
  Week 2, WBC, 3-5 | 1 | 3 | 2 | 3 | 1 | 3
  Week 2, WBC, 5-10 | 4 | 2 | 0 | 2 | 1 | 2
  Week 2, WBC, 10-15 | 0 | 0 | 0 | 1 | 0 | 0
  Week 2, WBC, 15-25 | 2 | 0 | 1 | 4 | 1 | 1
  Week 2, WBC, 25-50 | 3 | 3 | 4 | 2 | 9 | 2
  Week 2, WBC, 50-100 | 3 | 1 | 1 | 1 | 2 | 2
  Week 2, WBC, innumerable | 0 | 0 | 1 | 0 | 2 | 0
  Week 3, RBC, 0-1 | 3 | 0 | 1 | 0 | 1 | 1
  Week 3, RBC, 1-3 | 1 | 4 | 2 | 1 | 1 | 0
  Week 3, RBC, 3-5 | 0 | 0 | 0 | 0 | 0 | 0
  Week 3, RBC, 5-10 | 3 | 0 | 0 | 1 | 0 | 0
  Week 3, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 3, RBC, 15-25 | 0 | 1 | 0 | 0 | 0 | 0
  Week 3, RBC, 25-50 | 4 | 0 | 0 | 2 | 1 | 0
  Week 3, RBC, 50-100 | 0 | 1 | 0 | 1 | 0 | 0
  Week 3, RBC, innumerable | 0 | 0 | 0 | 0 | 1 | 0
  Week 3, WBC, 0-1 | 1 | 2 | 3 | 0 | 1 | 4
  Week 3, WBC, 1-3 | 4 | 1 | 2 | 1 | 1 | 3
  Week 3, WBC, 3-5 | 3 | 2 | 2 | 3 | 0 | 2
  Week 3, WBC, 5-10 | 4 | 4 | 2 | 3 | 1 | 2
  Week 3, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 3, WBC, 15-25 | 2 | 3 | 1 | 0 | 2 | 1
  Week 3, WBC, 25-50 | 2 | 1 | 1 | 2 | 3 | 2
  Week 3, WBC, 50-100 | 2 | 0 | 2 | 1 | 8 | 2
  Week 3, WBC, innumerable | 0 | 3 | 1 | 1 | 0 | 0
  Week 4, RBC, 0-1 | 1 | 0 | 0 | 0 | 4 | 1
  Week 4, RBC, 1-3 | 3 | 3 | 0 | 3 | 2 | 4
  Week 4, RBC, 3-5 | 1 | 0 | 0 | 1 | 1 | 0
  Week 4, RBC, 5-10 | 1 | 3 | 0 | 0 | 0 | 0
  Week 4, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4, RBC, 15-25 | 0 | 0 | 0 | 2 | 1 | 0
  Week 4, RBC, 25-50 | 0 | 0 | 1 | 1 | 1 | 1
  Week 4, RBC, 50-100 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4, RBC, innumerable | 1 | 0 | 0 | 0 | 0 | 0
  Week 4, WBC, 0-1 | 5 | 1 | 2 | 1 | 3 | 2
  Week 4, WBC, 1-3 | 5 | 2 | 1 | 4 | 4 | 1
  Week 4, WBC, 3-5 | 1 | 5 | 1 | 0 | 1 | 1
  Week 4, WBC, 5-10 | 2 | 1 | 0 | 2 | 4 | 3
  Week 4, WBC, 10-15 | 1 | 0 | 0 | 0 | 0 | 1
  Week 4, WBC, 15-25 | 0 | 3 | 3 | 3 | 4 | 2
  Week 4, WBC, 25-50 | 3 | 4 | 2 | 3 | 5 | 1
  Week 4, WBC, 50-100 | 2 | 1 | 1 | 1 | 1 | 1
  Week 4, WBC, innumerable | 1 | 1 | 0 | 1 | 2 | 0
  Week 6, RBC, 0-1 | 1 | 1 | 1 | 2 | 2 | 1
  Week 6, RBC, 1-3 | 1 | 4 | 1 | 2 | 2 | 2
  Week 6, RBC, 3-5 | 0 | 1 | 0 | 1 | 1 | 0
  Week 6, RBC, 5-10 | 0 | 1 | 0 | 1 | 1 | 0
  Week 6, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6, RBC, 15-25 | 1 | 0 | 1 | 0 | 1 | 1
  Week 6, RBC, 25-50 | 2 | 0 | 0 | 1 | 1 | 1
  Week 6, RBC, 50-100 | 1 | 0 | 0 | 0 | 0 | 0
  Week 6, RBC, innumerable | 0 | 0 | 0 | 0 | 0 | 0
  Week 6, WBC, 0-1 | 2 | 2 | 2 | 2 | 3 | 2
  Week 6, WBC, 1-3 | 4 | 5 | 6 | 4 | 3 | 1
  Week 6, WBC, 3-5 | 2 | 2 | 0 | 1 | 0 | 2
  Week 6, WBC, 5-10 | 0 | 2 | 0 | 2 | 1 | 1
  Week 6, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6, WBC, 15-25 | 2 | 1 | 2 | 1 | 4 | 2
  Week 6, WBC, 25-50 | 5 | 3 | 4 | 3 | 6 | 4
  Week 6, WBC, 50-100 | 2 | 2 | 1 | 1 | 1 | 1
  Week 6, WBC, innumerable | 3 | 1 | 0 | 1 | 2 | 0
  Week 8, RBC, 0-1 | 1 | 0 | 0 | 1 | 1 | 1
  Week 8, RBC, 1-3 | 1 | 5 | 1 | 2 | 2 | 1
  Week 8, RBC, 3-5 | 1 | 0 | 0 | 1 | 1 | 0
  Week 8, RBC, 5-10 | 0 | 1 | 0 | 1 | 0 | 0
  Week 8, RBC, 10-15 | 1 | 0 | 0 | 0 | 1 | 0
  Week 8, RBC, 15-25 | 2 | 1 | 0 | 0 | 1 | 0
  Week 8, RBC, 25-50 | 0 | 1 | 0 | 1 | 0 | 0
  Week 8, RBC, 50-100 | 1 | 0 | 0 | 1 | 0 | 0
  Week 8, RBC, innumerable | 0 | 0 | 0 | 0 | 1 | 0
  Week 8, WBC, 0-1 | 5 | 1 | 2 | 0 | 3 | 2
  Week 8, WBC, 1-3 | 5 | 0 | 1 | 4 | 6 | 3
  Week 8, WBC, 3-5 | 0 | 1 | 2 | 3 | 3 | 0
  Week 8, WBC, 5-10 | 3 | 3 | 1 | 2 | 1 | 0
  Week 8, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 1
  Week 8, WBC, 15-25 | 0 | 2 | 2 | 2 | 5 | 1
  Week 8, WBC, 25-50 | 1 | 0 | 2 | 4 | 3 | 1
  Week 8, WBC, 50-100 | 3 | 1 | 2 | 0 | 3 | 1
  Week 8, WBC, innumerable | 2 | 0 | 0 | 0 | 2 | 1
  Week 12, RBC, 0-1 | 1 | 1 | 1 | 0 | 1 | 0
  Week 12, RBC, 1-3 | 1 | 2 | 5 | 2 | 3 | 1
  Week 12, RBC, 3-5 | 0 | 0 | 0 | 0 | 0 | 1
  Week 12, RBC, 5-10 | 1 | 1 | 1 | 1 | 0 | 0
  Week 12, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12, RBC, 15-25 | 2 | 0 | 0 | 1 | 1 | 0
  Week 12, RBC, 25-50 | 0 | 0 | 1 | 1 | 0 | 0
  Week 12, RBC, 50-100 | 2 | 0 | 0 | 0 | 1 | 0
  Week 12, RBC, innumerable | 0 | 0 | 0 | 0 | 0 | 0
  Week 12, WBC, 0-1 | 2 | 3 | 4 | 3 | 3 | 1
  Week 12, WBC, 1-3 | 6 | 2 | 2 | 0 | 3 | 4
  Week 12, WBC, 3-5 | 2 | 0 | 1 | 1 | 0 | 1
  Week 12, WBC, 5-10 | 2 | 1 | 2 | 3 | 1 | 0
  Week 12, WBC, 10-15 | 0 | 0 | 0 | 1 | 0 | 0
  Week 12, WBC, 15-25 | 2 | 2 | 2 | 0 | 2 | 1
  Week 12, WBC, 25-50 | 3 | 5 | 2 | 1 | 2 | 3
  Week 12, WBC, 50-100 | 4 | 0 | 1 | 3 | 4 | 0
  Week 12, WBC, innumerable | 1 | 0 | 1 | 1 | 1 | 1
  Week 13, RBC, 0-1 | 2 | 0 | 0 | 1 | 1 | 0
  Week 13, RBC, 1-3 | 2 | 5 | 2 | 2 | 3 | 1
  Week 13, RBC, 3-5 | 1 | 0 | 0 | 0 | 0 | 1
  Week 13, RBC, 5-10 | 1 | 1 | 0 | 1 | 1 | 0
  Week 13, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 13, RBC, 15-25 | 2 | 0 | 0 | 0 | 0 | 2
  Week 13, RBC, 25-50 | 0 | 0 | 0 | 0 | 0 | 0
  Week 13, RBC, 50-100 | 1 | 0 | 0 | 1 | 0 | 0
  Week 13, RBC, innumerable | 0 | 0 | 0 | 0 | 0 | 0
  Week 13, WBC, 0-1 | 4 | 1 | 1 | 1 | 2 | 0
  Week 13, WBC, 1-3 | 0 | 4 | 2 | 5 | 2 | 2
  Week 13, WBC, 3-5 | 3 | 2 | 2 | 1 | 6 | 1
  Week 13, WBC, 5-10 | 1 | 1 | 1 | 0 | 2 | 0
  Week 13, WBC, 10-15 | 0 | 0 | 0 | 1 | 0 | 0
  Week 13, WBC, 15-25 | 1 | 3 | 0 | 1 | 3 | 2
  Week 13, WBC, 25-50 | 2 | 1 | 3 | 1 | 4 | 3
  Week 13, WBC, 50-100 | 3 | 0 | 1 | 3 | 1 | 0
  Week 13, WBC, innumerable | 0 | 1 | 0 | 0 | 1 | 0
  Week 14, RBC, 0-1 | 0 | 0 | 0 | 0 | 0 | 1
  Week 14, RBC, 1-3 | 5 | 5 | 4 | 2 | 2 | 1
  Week 14, RBC, 3-5 | 0 | 0 | 0 | 0 | 1 | 0
  Week 14, RBC, 5-10 | 1 | 1 | 1 | 0 | 0 | 1
  Week 14, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14, RBC, 15-25 | 0 | 0 | 0 | 1 | 0 | 1
  Week 14, RBC, 25-50 | 1 | 1 | 0 | 1 | 1 | 0
  Week 14, RBC, 50-100 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14, RBC, innumerable | 0 | 0 | 0 | 1 | 0 | 0
  Week 14, WBC, 0-1 | 3 | 1 | 1 | 2 | 2 | 3
  Week 14, WBC, 1-3 | 0 | 1 | 3 | 5 | 2 | 1
  Week 14, WBC, 3-5 | 1 | 1 | 1 | 0 | 0 | 1
  Week 14, WBC, 5-10 | 1 | 1 | 0 | 3 | 1 | 1
  Week 14, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14, WBC, 15-25 | 2 | 2 | 2 | 2 | 4 | 1
  Week 14, WBC, 25-50 | 4 | 3 | 3 | 2 | 3 | 3
  Week 14, WBC, 50-100 | 1 | 1 | 0 | 2 | 3 | 0
  Week 14, WBC, innumerable | 2 | 1 | 0 | 0 | 1 | 0
  Week 15, RBC, 0-1 | 2 | 0 | 1 | 1 | 0 | 0
  Week 15, RBC, 1-3 | 2 | 4 | 1 | 0 | 5 | 1
  Week 15, RBC, 3-5 | 1 | 0 | 0 | 2 | 0 | 1
  Week 15, RBC, 5-10 | 4 | 0 | 0 | 0 | 0 | 0
  Week 15, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 15, RBC, 15-25 | 0 | 2 | 0 | 2 | 0 | 0
  Week 15, RBC, 25-50 | 0 | 1 | 0 | 1 | 0 | 0
  Week 15, RBC, 50-100 | 1 | 0 | 0 | 1 | 1 | 0
  Week 15, RBC, innumerable | 0 | 0 | 1 | 1 | 2 | 0
  Week 15, WBC, 0-1 | 1 | 1 | 1 | 1 | 1 | 1
  Week 15, WBC, 1-3 | 5 | 3 | 3 | 1 | 3 | 0
  Week 15, WBC, 3-5 | 2 | 0 | 0 | 3 | 2 | 1
  Week 15, WBC, 5-10 | 2 | 0 | 1 | 1 | 1 | 0
  Week 15, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 15, WBC, 15-25 | 3 | 1 | 2 | 2 | 2 | 4
  Week 15, WBC, 25-50 | 1 | 0 | 2 | 3 | 2 | 3
  Week 15, WBC, 50-100 | 2 | 2 | 2 | 1 | 1 | 0
  Week 15, WBC, innumerable | 1 | 1 | 0 | 0 | 4 | 0
  Week 16, RBC, 0-1 | 1 | 0 | 0 | 0 | 1 | 1
  Week 16, RBC, 1-3 | 4 | 5 | 1 | 3 | 2 | 1
  Week 16, RBC, 3-5 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16, RBC, 5-10 | 0 | 2 | 0 | 0 | 0 | 1
  Week 16, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16, RBC, 15-25 | 0 | 2 | 0 | 0 | 0 | 1
  Week 16, RBC, 25-50 | 0 | 2 | 0 | 1 | 0 | 0
  Week 16, RBC, 50-100 | 1 | 0 | 0 | 0 | 1 | 0
  Week 16, RBC, innumerable | 1 | 0 | 0 | 0 | 0 | 1
  Week 16, WBC, 0-1 | 1 | 0 | 1 | 2 | 3 | 1
  Week 16, WBC, 1-3 | 1 | 2 | 1 | 3 | 4 | 3
  Week 16, WBC, 3-5 | 1 | 1 | 0 | 1 | 1 | 1
  Week 16, WBC, 5-10 | 0 | 1 | 0 | 1 | 1 | 1
  Week 16, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16, WBC, 15-25 | 1 | 2 | 3 | 0 | 2 | 3
  Week 16, WBC, 25-50 | 5 | 5 | 3 | 5 | 4 | 2
  Week 16, WBC, 50-100 | 0 | 0 | 1 | 1 | 1 | 1
  Week 16, WBC, innumerable | 1 | 1 | 1 | 1 | 0 | 0
  Week 20, RBC, 0-1 | 1 | 0 | 1 | 1 | 3 | 1
  Week 20, RBC, 1-3 | 2 | 5 | 4 | 1 | 4 | 2
  Week 20, RBC, 3-5 | 0 | 0 | 0 | 1 | 0 | 0
  Week 20, RBC, 5-10 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20, RBC, 15-25 | 1 | 0 | 0 | 0 | 1 | 0
  Week 20, RBC, 25-50 | 0 | 1 | 0 | 0 | 0 | 0
  Week 20, RBC, 50-100 | 2 | 0 | 0 | 1 | 0 | 0
  Week 20, RBC, innumerable | 1 | 0 | 0 | 0 | 0 | 0
  Week 20, WBC, 0-1 | 4 | 0 | 1 | 1 | 4 | 1
  Week 20, WBC, 1-3 | 2 | 1 | 3 | 2 | 2 | 3
  Week 20, WBC, 3-5 | 2 | 2 | 1 | 0 | 3 | 0
  Week 20, WBC, 5-10 | 2 | 0 | 0 | 1 | 0 | 2
  Week 20, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20, WBC, 15-25 | 0 | 0 | 2 | 1 | 1 | 2
  Week 20, WBC, 25-50 | 2 | 3 | 1 | 5 | 6 | 1
  Week 20, WBC, 50-100 | 2 | 2 | 1 | 0 | 3 | 0
  Week 20, WBC, innumerable | 2 | 0 | 0 | 0 | 2 | 1
  Week 24, RBC, 0-1 | 2 | 0 | 0 | 1 | 0 | 0
  Week 24, RBC, 1-3 | 4 | 6 | 1 | 0 | 4 | 2
  Week 24, RBC, 3-5 | 0 | 0 | 0 | 0 | 0 | 2
  Week 24, RBC, 5-10 | 0 | 0 | 0 | 0 | 0 | 1
  Week 24, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24, RBC, 15-25 | 2 | 0 | 1 | 1 | 1 | 0
  Week 24, RBC, 25-50 | 1 | 0 | 1 | 0 | 4 | 0
  Week 24, RBC, 50-100 | 1 | 0 | 1 | 1 | 0 | 0
  Week 24, RBC, innumerable | 0 | 0 | 0 | 0 | 0 | 0
  Week 24, WBC, 0-1 | 5 | 2 | 0 | 1 | 1 | 2
  Week 24, WBC, 1-3 | 2 | 4 | 2 | 3 | 5 | 1
  Week 24, WBC, 3-5 | 1 | 2 | 1 | 0 | 2 | 3
  Week 24, WBC, 5-10 | 0 | 0 | 1 | 2 | 1 | 1
  Week 24, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24, WBC, 15-25 | 2 | 2 | 0 | 1 | 2 | 0
  Week 24, WBC, 25-50 | 2 | 4 | 4 | 3 | 4 | 2
  Week 24, WBC, 50-100 | 3 | 2 | 1 | 0 | 2 | 1
  Week 24, WBC, innumerable | 0 | 1 | 1 | 1 | 2 | 0
  Week 25, RBC, 0-1 | 0 | 1 | 1 | 1 | 0 | 0
  Week 25, RBC, 1-3 | 2 | 1 | 0 | 3 | 3 | 3
  Week 25, RBC, 3-5 | 0 | 2 | 1 | 0 | 2 | 0
  Week 25, RBC, 5-10 | 1 | 1 | 0 | 0 | 0 | 0
  Week 25, RBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 25, RBC, 15-25 | 1 | 1 | 2 | 0 | 1 | 1
  Week 25, RBC, 25-50 | 0 | 0 | 1 | 1 | 0 | 0
  Week 25, RBC, 50-100 | 1 | 0 | 0 | 0 | 0 | 0
  Week 25, RBC, innumerable | 0 | 0 | 2 | 0 | 0 | 0
  Week 25, WBC, 0-1 | 1 | 3 | 3 | 1 | 2 | 1
  Week 25, WBC, 1-3 | 1 | 0 | 0 | 0 | 6 | 0
  Week 25, WBC, 3-5 | 2 | 0 | 2 | 2 | 1 | 0
  Week 25, WBC, 5-10 | 0 | 3 | 1 | 2 | 0 | 2
  Week 25, WBC, 10-15 | 0 | 0 | 0 | 0 | 0 | 0
  Week 25, WBC, 15-25 | 4 | 0 | 1 | 2 | 2 | 1
  Week 25, WBC, 25-50 | 1 | 3 | 2 | 1 | 4 | 3
  Week 25, WBC, 50-100 | 3 | 0 | 2 | 1 | 1 | 0
  Week 25, WBC, innumerable | 0 | 1 | 1 | 0 | 1 | 0

26. Secondary Outcome: Population Pharmacokinetic (PK) Parameter of Plasma Concentration of DEN
Description: A total of 6 blood samples, 2 milliliter each were planned to be obtained over the course of the study for determination of DEN plasma concentrations. For each PK sampling visit a sampling interval was defined. PK samples were planned to be collected at any time during the defined sampling intervals.
Time Frame: Pre-dose at Week 0, 0.5 to 1.5 h post-dose at Week 4, 12, 16 or 20, 2 to 4 h post-dose at Week 4, 12, 16 or 20 and 6 to 10 h post-dose at Week 4, 12, 16 or 20
Population: Sparse PK (PPK) Population comprised of all those participants who were assigned to the sparse (population PK) group. All consenting participants were eligible for inclusion in the sparse PK population except for those participants participating in the serial PK assessment. The data for this outcome measure was not collected.
Arm/Group | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Descriptive Statistics of Dipeptidyl Peptidase-IV (DPP-IV) Inhibition Performed as Part of the Population PK
Description: A total of 6 blood samples, 2 milliliter each were planned to be obtained over the course of the study for determination of DPP-IV inhibition. For each PK sampling visit a sampling interval was defined. PK samples were planned to be collected at any time during the defined sampling intervals.
Time Frame: as for outcome 26
Population: PPK Population. The data for this outcome measure was not collected.
Groups:
- DEN 7.5 mg: Participants received oral dose of DEN 2.5 mg capsule once daily in the morning, 30 min prior to breakfast during the main phase/extension phase 12-weeks treatment period. Participants were dispensed 3 bottles (bottle A, B and C) and were instructed to take 1 capsule daily from each bottle such that taking 1 capsule from each bottle daily provided the appropriate dose of DEN 2.5 mg to the participants.
Arm/Group | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's were collected up to Follow-up (up to Week 25)
Description: Safety Population was used.
Arm/Group | Placebo | DEN 2.5 mg | DEN 7.5 mg | DEN 15 mg | DEN 30 mg | DEN 45 mg
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/61 | 0/63 | 0/66 | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/64 | 1/61 | 2/63 | 0/66 | 4/60 | 3/61
Other Adverse Events (participants affected / at risk) | 6/64 | 5/61 | 8/63 | 11/66 | 6/60 | 3/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | DEN 2.5 mg (N=61) | DEN 7.5 mg (N=63) | DEN 15 mg (N=66) | DEN 30 mg (N=60) | DEN 45 mg (N=61)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | DEN 2.5 mg (N=61) | DEN 7.5 mg (N=63) | DEN 15 mg (N=66) | DEN 30 mg (N=60) | DEN 45 mg (N=61)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 7 | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.